CLINICAL TRIAL: NCT05812417
Title: An Open-label, Single-dose, Parallel-group Study to Evaluate the Effects of Renal Function on Pharmacokinetics and Safety of DA-8010
Brief Title: A Study to Evaluate the Effects of Renal Function on Pharmacokinetics and Safety of DA-8010
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DA8010_RI_I
Record Dates: First submitted 2023-03-20; First posted 2023-04-13 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Renal Impairment; Healthy
MeSH Terms: conditions — Renal Insufficiency | interventions — DA-8010

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal renal function (Active Comparator): eGFR >=90 mL/min/1.73m^2
  Interventions: Drug: DA-8010
- Mild renal impairment (Experimental): eGFR 60~89 mL/min/1.73m^2
  Interventions: Drug: DA-8010
- Moderate renal impairment (Experimental): eGFR 30~59 mL/min/1.73m^2
  Interventions: Drug: DA-8010
- Severe renal impairment (Experimental): eGFR 15~29 mL/min/1.73m^2
  Interventions: Drug: DA-8010

INTERVENTIONS:
Drug: DA-8010 — DA-8010 5mg single dose administration

SUMMARY:
This Study will evaluate the effects of renal function on pharmacokinetics and safety of DA-8010

ELIGIBILITY:
Inclusion Criteria:

[Healthy Volunteer]

* Adult male or female, 19 years to 75 years
* eGFR ≥ 90 mL/min/1.73m^2
* Body weight over 45.0 kg and body mass index in the range of 18.0 to 40.0 kg/m^2
* The subjects signed and dated informed consent form after hearing a detailed explanation of the study, fully understanding and determined voluntarily to participate
* The subjects who are judged appropriate to participate this clinical trial according to the physical examination, laboratory examination and questionnaire

[Renal Impairment Patient]

* Adult male of female, 19 years to 75 years
* eGFR < 90 mL/min/1.73m^2, not on dialysis
* Body weight over 45.0 kg and body mass index in the range of 18.0 to 40.0kg/m^2
* The subjects signed and dated informed consent form after hearing a detailed explanation of the study, fully understanding and determined voluntarily to participate
* The subjects who are judged appropriate to participate this clinical trial according to the physical examination, laboratory examination and questionnaire

Exclusion Criteria:

* The subjects with acute illness
* The subjects with a history of gastrointestinal disease or surgery that may affect the absorption of Investigational Product
* The subjects hypersensitive to any of the Investigational Product components or other drug components
* The subjects who have continuously consumed excessive smoking or alcohol within 6 months of screening, or who cannot stop smoking, caffeine, or alcohol intake during hospitalization
* The subjects who have history of drug abuse
* The subjects who are pregnant or lactating
* The subjects who do not agree to exclude the possibility of pregnancy using the contraception from the date of the first administration of the Investigational Product until the 4 weeks after the last administration

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve over the time interval from 0 to the last quantifiable plasma concentration (AUClast) of DA-8010 | Pre-dose, 1hour, 2hour, 3hour, 3.5hour, 4hour, 4.5hour, 5hour, 5.5hour, 6hour, 6.5hour, 7hour, 8hour, 12hour, 24hour, 48hour post-dosing on Day 1
Peak Plasma Concentration (Cmax) of DA-8010 | Pre-dose, 1hour, 2hour, 3hour, 3.5hour, 4hour, 4.5hour, 5hour, 5.5hour, 6hour, 6.5hour, 7hour, 8hour, 12hour, 24hour, 48hour post-dosing on Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Bundang Medical Center, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes